CLINICAL TRIAL: NCT02298218
Title: Clinical Study About the Role of COX-2 Inhibitor in Liver Cirrhosis With Biliary Atresia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0597
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Biliary Atresia, Kasai Portoenterostomy Status
MeSH Terms: conditions — Biliary Atresia | interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meloxicam (Experimental): The intervention drug, meloxicam is safe medicine which is used to treat pain or inflammation caused by osteoarthritis or rheumatoid arthritis in adults and children who are at least 2 years old. It may also be used for purposes not listed in the medication guide. It will be taken once a daily with a dose of 0.125 mg/kg/day (high-dose group) or 0.06 mg/kg/day (low-dose group). After 6 months of medication, the maintenance will be decided by the comparison of liver stiffness score before and after the intervention.
  Interventions: Drug: Meloxicam
- No intervention (No Intervention): During 6 months, without meloxicam, the maintenance will be decided by the comparison of liver stiffness score comparing the intervention group.

INTERVENTIONS:
Drug: Meloxicam — The intervention drug, meloxicam is safe medicine which is used to treat pain or inflammation caused by osteoarthritis or rheumatoid arthritis in adults and children who are at least 2 years old. It may also be used for purposes not listed in the medication guide. It will be taken once a daily with a dose of 0.125 mg/kg/day (high-dose group) or 0.06 mg/kg/day (low-dose group). After 6 months of medication, the maintenance will be decided by the comparison of liver stiffness score before and after the intervention.
  Arms: Meloxicam

SUMMARY:
In this clinical study, meloxicam will be used to the patients who are older than 2 years and underwent Kasai portoenterostomy to treat their biliary atresia before. Before and after the medication, their liver stiffness scores will be checked using hepatic Fibroscan. Liver stiffness scores will be compared before and after the medication of meloxicam, and the roll of the COX-2 inhibitor (meloxicam) in the patients with biliary atresia in releasing their hepatic fibrosis. Also, the side effect of the drug will be checked. The intervention drug, meloxicam is safe medicine which is used to treat pain or inflammation caused by osteoarthritis or rheumatoid arthritis in adults and children who are at least 2 years old. It may also be used for purposes not listed in the medication guide. It will be taken once a daily with a dose of 0.125 mg/kg/day (high-dose group) or 0.06 mg/kg/day (low-dose group). After 6 months of medication, the maintenance will be decided by the comparison of liver stiffness score before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had undergone a Kasai portoenterostomy for BA, and who were postoperatively managed in our outpatient clinic
2. Patients who made informed consent for clinical study of COX-2 inhibitor
3. Patients who were followed up with liver fibroscan study
4. Patients who were over 2 years old and less than or equal to 17 years

Exclusion Criteria:

1. Patients who were impossible to join the clinical study because of their underlying diseases (renal disease, liver disease, diabetes mellitus, GI disease, including bleeding, perforation, or ulceration, etc.) other than biliary atresia, ii) H. pylori infection, iii) asthma, iv) nasal polyp, v) hypertension, vi) hematologic disease, vii) coagulopathy, viii) cardiac disease, ix) vascular disease
2. Patients who did not get the drug (COX-2 inhibitor)
3. Patients who did not check liver fibroscan
4. Patients who were impossible to join the clinical study because of their complication after Kasai portoenterostomy
5. Patients who did not make informed consent for clinical study of COX-2 inhibitor
6. Patients who cannot take drug because of their allergy, skin disease or asthma attack to drug (COX-2 inhibitor)
7. Patients who were decided to withdraw because of their severe drug adverse events

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
liver stiffness score on FibroScan | from 6 to 12 years
  statistical comparison between liver stiffness score of study group (COX-2 inhibitor group) and control group (no intervention group) before and after the clinical study using t-test, chi-square and logistic regression test)

CONTACTS AND LOCATIONS:
Overall Officials: Seok Joo Han, MD, Principal Investigator — Department of Pediatric Surgery, Severance Children's Hospital, Yonsei University College of Medicine